CLINICAL TRIAL: NCT04102813
Title: Neurobiological and Anti-inflammatory Effects of a Deep Diaphragmatic Breathing Technique Based on Functional Psychotherapy: a Randomised Clinical Trial
Brief Title: Deep Diaphragmatic Breathing: Neurobiological and Anti-inflammatory Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other)
Collaborators: Centro Studi Psicoterapia Neo-Funzionale (Unknown)
Responsible Party: Principal Investigator, Giuseppe Maniaci, Adjunct Professor, Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06/2019
Record Dates: First submitted 2019-09-19; First posted 2019-09-25 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Unrecognized Condition
Keywords: deep diaphragmatic breathing; cortisol; sympathetic nervous system; parasympathetic nervous system; inflammatory cytokines; Functional psychotherapy

STUDY DESIGN:
Intervention Model Description: After a psychiatric, psychological and anthropometric assessment, healthy volunteers will receive the Trier Social Stress Test (TSST) procedure and than they are randomly assigned to 30 min of deep diagrammatic breathing based on Functional therapy (FT) or attention control (AC). All subjects are tested at the baseline (T0), at the end of the TSST (T1), at the end of the treatment (T2) and 30 minutes after the treatment (T3)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects are advised that they are going to receive some kind of psychological support after a psychosocial stress. The investigator isn't informed about the randomisation procedures of the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Therapy (FT) (Experimental): The FT includes a variety of functional techniques such as diaphragmatic breathing, and thoracic and abdominal manipulation, designed to stimulate the neurofunctional interconnection between body, mind and immune system. The FT session will last 30 minutes.
  Interventions: Behavioral: Functional Therapy
- Attention Control (AC) (No Intervention): The AC group will listen an audiobook lasting for 30 minutes, which will be used as attention control activity

INTERVENTIONS:
Behavioral: Functional Therapy — It consists in a group of body-mind techniques based on functional theory developed in Italy by prof. Luciano Rispoli. These techniques are oriented to stimulate a diaphragmatic breathing though a thoracic and abdominal manipulation, with the aim to activate the parasympathetic nervous system and therefore reducing inflammation
  Arms: Functional Therapy (FT)

SUMMARY:
The exposure to acute and\or chronic stress can produce an activation of sympathetic nervous system (SNS), leading to an increased level of cortisol and pro-inflammatory cytokines. The mind-body techniques (MBT), such as diaphragmatic breathing, mindfulness, and Yoga, have demonstrated their validity in reducing mental stress and relieving inflammatory conditions. The aim of our study is to verify the efficacy of a single Functional Therapy (FT) session to relieve inflammations, decreasing cortisol levels and activating the parasympathetic nervous system in healthy subjects after the administration of an acute stress such as the Trier Social Stress Test (TSST) protocol. After a psychiatric, psychological and anthropometric assessment, participants are randomly assigned to FT or attention placebo control group. The FT session lasting for 30 minutes and is conducted by therapists specialized in the MBT. The treatment's efficacy in reducing inflammatory states is verified by measuring the variations of the hearth rate, skin conductance, electromyography, pro-inflammatory cytokines (IL-6, TNFα, IL1β), anti-inflammatory cytokine (IL-10), and salivary cortisol; furthermore, the State Trait Anxiety Inventory (STAI) (state and trait) and Subjective Units of Distress Scale (SUDS) questionnaires are used as psychometric measures of anxiety and stress. All the participants are tested at baseline, at the end of TSST, at the end of the FT or audiobook session, and at follow-up 30 minutes after the session.

DETAILED DESCRIPTION:
Life's dynamics in modern societies expose the individuals to high level of suffering and stress, which can affect both psychological and physiological well-being. Numerous scientific evidences showed the correlation between stress and immunity system dysregulation. The exposure to acute and\or chronic mental stress conditions can alter the physiological functions of the organism, through the activation of sympathetic nervous system (SNS) and the inhibition of the parasympathetic nervous system (PNS). The activation of peripheral and central immune-inflammatory pathways is indicated by increased levels of proinflammatory cytokines, such as Interleukin-1 β (IL-1β), Interleukin-6 (IL-6), and Tumor necrosis factor-α (TNFα). Furthermore, experiencing high stress levels may lead to a disruption of the Hypothalamic-Pituitary-Adrenal (HPA) axis, with consequent increasing of cortisol's level, low-grade systemic inflammation and oxidative stress. These results correlate with the develop and progression of a wide range of pathological conditions, such as cardiovascular disease, Type II diabetes, arthritis, osteoporosis, Alzheimer's disease, and depression. In addition, inflammation is now considered as a risk factor for most cancers' disease, promoting pathological mechanism such as proliferation, angiogenesis and metastases.

The last 20 years has seen an exponential growth of the mind-body techniques (MBT), an heterogeneous group of exercises and techniques focusing the life-styles, which has demonstrated validity in the reduction of psychological stress and inflammatory states. The techniques adopted by the clinical trials available include Yoga, Mindfulness, Tai Chi Chih, and Qigong; these protocols last usually from 4 to 12 weeks, and have been applied on clinical samples ranging on heterogeneous pathological conditions. However, the techniques used in the majority of these studies are derived from eastern meditative tradition and were not primarily developed to carrying out anti-inflammatory effects. Furthermore, the data concerning the effects of a single session of MBT under controlled experimental conditions are still lacking. In this regard, the Functional Therapy (FT) approach, an integrated body-mind therapy developed around the knowledges of psychoneuroimmunology (PNI), represents a potentially effective and specific methodology to counteract the physiological and psychological effects caused by prolonged exposure to stress conditions.

Given these premises, the aim of this clinical trial is to verify the efficacy of a single Functional Therapy (FT) session to relieve inflammations, decreasing cortisol levels and activating the parasympathetic nervous system in healthy subjects after the administration of an acute stress such as the Trier Social Stress Test (TSST).

Patients will be recruited starting in October 2019, via advertisement posted in university classrooms and premises. Researchers planned to recruit a sample of 40 participants. For the recruitment a structured telephone screening will help the researchers to investigate on some exclusion criteria. Then a consultation with a clinical psychologist and a psychiatrist will be programmed together with the administration of the psychological tests. Psychological assessment includes an ad-hoc sociodemographic questionnaire; a shortened version of Wechsler Adult Intelligence Scale - Revised (WAIS-R); Millon Clinical Multiaxial Inventory-III (MCMI-III); and Stress-related Vulnerability Scale (SVS). All these assessments will take place in the outpatient clinic of the policlinic "P. Giaccone", Palermo. After the assessment, eligible subjects will be randomized in the FT group or in the attention control group (AC), and will be assigned to the next therapist on a time capacity list.

All the sessions will be taking place in the Neo-Functional Psychotherapy Centre of Palermo. During the session, participants will be assessed for anthropometric, psychological, biofeedback and salivary parameters. Anthropometric parameters include height, weight, and BMI; Psychological assessment includes the State-Trait Anxiety Inventory, in both trait and state form; and Subjective Unit of Distress Scale. Biofeedback parameters include hearth rate, skin conductance, and electromyography. Salivary measurements include pro-inflammatory cytokines (IL-6, TNFα, IL1β), anti-inflammatory cytokine (IL-10), and cortisol.

Upon arrival, the anthropometric parameters will be assessed, thus biofeedback sensors will be connected to participants and it will record, for 5 minutes, the physiological parameters that will constitute the baseline; biofeedback sensors will remain online for the whole duration of the clinical trial. During this phase the STAI (trait and state) and SUDS questionnaires will be administered, and the first salivary samples will be taken for cortisol and cytokines.

Then, participants will be submitted to the TSST social stress, a protocol used by researchers to induce stress under controlled condition. TSST is divided in 5 minutes components and the whole procedure lasts approximately 15 minutes; at the end, the second psychological and salivary assessments will be carried out.

Participants will be randomized in FT group or AC group. Five different therapists with a 4-year postgraduate training on functional approach will apply the FT session. The treatment was specifically manualized to reducing stress condition and to relieve inflammatory states. Specifically, the treatment includes a variety of functional techniques such as diaphragmatic breathing, and thoracic and abdominal manipulation, designed to stimulate the neurofunctional interconnection between body, mind and immune system. The FT session will last 30 minutes. The participants assigned to the AC will listen an audiobook lasting for 30 minutes, which will be used as attention placebo control activity. At the end of the session, the third psychological and salivary assessments will be carried out.

Finally, all the participants will be undergoing to a follow-up phase, designed to assess the biofeedback and cytokines slow-responses to stress and relaxation procedures. Thus, subjects will be provided with an additionally 30 minutes session of audiobook listening, used as attention control placebo. At the end of the session, the fourth psychological and salivary assessments will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aging between 18 and 55;
* Able to understanding and signing the informed consent;

Exclusion Criteria:

* a current or lifetime diagnosis of any psychiatric disorders
* a past or present of drug abuse or drug addiction (including nicotine)
* chronic inflammation diseases
* Taking medicines active on the immune system (antibiotics, anti-histamines, corticosteroids, psychotropic substances) during the 2 weeks prior to the operation;
* Intense physical activities (at least 1h\day);
* Intelligence Quotient less than 65
* BMI more than 40
* serious infections (such as HIV, hepatitis B and C)
* cancer in the previous 6 months
* regular use of anti-inflammatory drugs for more than 15 days/month
* Participation to other clinical trials;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Heart rate values measured by biofeedback sensor | end of the treatment after the TSST (30 minutes) and 30 minutes later (follow-up)
  change of heart rate values indicating a relaxation state (measured by blood volume pulse). Higher values of heart rate represent worst parasympathetic activity
Skin conductance values measured by biofeedback sensor | end of the treatment after the TSST (30 minutes) and 30 minutes later (follow-up)
  change of skin conductance values indicating a relaxation state (measured through micro-Siemens). Lower values of skin conductance represent worst parasympathetic activity
Surface electromyography values measured by biofeedback sensor on left deltoid | end of the treatment after the TSST (30 minutes) and 30 minutes later (follow-up)
  change of Electromyography values indicating a relaxation state (measured through microvolts). Higher values of skin conductance represent worst parasympathetic activity
cortisol levels measured by saliva sample | end of the treatment after the TSST (30 minutes) and 30 minutes later (follow-up)
  change of cortisol levels measured by ng/ml. Higher values indicate worst stress levels
inflammation parameters measured by saliva sample | end of the treatment after the TSST (30 minutes) and 30 minutes later (follow-up)
  change of pro-inflammatory (IL-6, TNFα, IL1β), and of anti-inflammatory (IL-10) cytokines measured by pg/mL. Higher levels of IL-6, TNFα, IL1β and lower levels of IL-10 indicate an inflammation
state anxiety measured by State Trait Anxiety Inventory | end of the treatment after the TSST (30 minutes) and 30 minutes later (follow-up)
  change of state anxiety (measured by State Trait Anxiety Inventory questionnaire). The score is from 20 to 80. Higher values indicate a worst state anxiety
perceived stress measured by Subjective Units of Distress Scale | end of the treatment after the TSST (30 minutes) and 30 minutes later (follow-up)
  change of perceived stress (measured by Subjective Units of Distress Scale questionnaire).The score is from 0 to 10. Higher values indicate a worst perceived stress

CONTACTS AND LOCATIONS:
Locations (1):
- Unit of Psychiatry, Palermo, PA, Italy

REFERENCES:
- [Derived] Maniaci G, Daino M, Iapichino M, Giammanco A, Taormina C, Bonura G, Sardella Z, Carolla G, Cammareri P, Sberna E, Clesi MF, Ferraro L, Gambino CM, Ciaccio M, Rispoli L, La Cascia C, La Barbera D, Quattrone D. Neurobiological and Anti-Inflammatory Effects of a Deep Diaphragmatic Breathing Technique Based on Neofunctional Psychotherapy: A Pilot RCT. Stress Health. 2024 Dec;40(6):e3503. doi: 10.1002/smi.3503. Epub 2024 Nov 14. PMID 39543797